CLINICAL TRIAL: NCT07246876
Title: Diagnostic Value of EBUS-Guided Transbronchial Mediastinal Cryobiopsy Versus Conventional Bronchoscopic Approaches for Stage I/II Sarcoidosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Principal Investigator, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DETECTION-SAR-II
Record Dates: First submitted 2025-11-19; First posted 2025-11-24 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Sarcoidosis, Pulmonary
Keywords: Endobronchial Ultrasound; EBUS-TBNA; EBUS-transbronchial mediastinal cryobiopsy; Sarcoidosis
MeSH Terms: conditions — Sarcoidosis, Pulmonary; Sarcoidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EBUS-TBMC (Experimental): Patients will receive endobronchial biopsy, transbronchial lung biopsy and EBUS-TBMC
  Interventions: Procedure: EBUS-TBMC based sampling method
- EBUS-TBNA (Experimental): Patients will receive endobronchial biopsy, transbronchial lung biopsy and EBUS-TBNA
  Interventions: Procedure: EBUS-TBNA-based sampling methods

INTERVENTIONS:
Procedure: EBUS-TBNA-based sampling methods — Participants will receive an endobronchial biopsy and a transbronchial lung biopsy, followed by EBUS-TBNA.
  Arms: EBUS-TBNA
Procedure: EBUS-TBMC based sampling method — Participants will receive an endobronchial biopsy and a transbronchial lung biopsy, followed by EBUS-TBMC.
  Arms: EBUS-TBMC

SUMMARY:
Endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA), combined with endobronchial biopsy (EBB) and/or transbronchial lung biopsy (TBLB), and endobronchial ultrasound-guided transbronchial mediastinal cryobiopsy (EBUS-TBMC) have high diagnostic yields for patients with sarcoidosis. However, a direct comparison between them has not been conducted. This randomized controlled trial aims to compare directly the diagnostic yield between EBUS-TBMC and EBUS-TBNA+EBB+TBLB in sarcoidosis.

DETAILED DESCRIPTION:
Endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA), combined with endobronchial biopsy (EBB) and/or transbronchial lung biopsy (TBLB), and endobronchial ultrasound-guided transbronchial mediastinal cryobiopsy (EBUS-TBMC) have high diagnostic yields for patients with sarcoidosis. However, a direct comparison between them has not been conducted. Two questions remain need to be answered: (1) Does EBUS-TBMC have the same or better diagnostic sensitivity for sarcoidosis than EBUS-TBNA combined with standard bronchoscopic modalities (EBB or/and TBLB)? (2) Can combining EBUS-TBMC with standard bronchoscopic modalities further increase the diagnostic sensitivity for sarcoidosis? This study is designed as a randomised controlled trial to compare the diagnostic yield between EBUS-TBMC and conventional bronchoscopic approaches for diagnosing stage I/II sarcoidosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18years;
2. Patients with clinical and radiological suspicion of stage I or stage II sarcoidosis;
3. Fully informed of the purpose and method of the study

Exclusion Criteria:

1. Pathologically confirmed sarcoidosis, obvious organ involvement with the possibility of confirming granulomas using a minimally invasive diagnostic procedure;
2. Patients with medical contraindications to bronchoscopy procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 469 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The granuloma detection rate | 7 days after sampling
  The number of patients with granulomas detected relative to the total number of patients tested.

SECONDARY OUTCOMES:
Diagnostic yield | 6 Month after sampling
  The proportion of all participants who underwent the diagnostic procedure in whom a specific malignant or benign diagnosis was established
Negative predictive value | 6 months after sampling
Incidence of complications | 4 weeks after sampling